CLINICAL TRIAL: NCT06416709
Title: To Study the Clinical Treatment Plan of Lung Injury Caused by Major Infectious Diseases Treated With Stem Cells
Brief Title: Stem Cell Treatment for Lung Injury Caused by Major Infectious Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cell Energy Life Sciences Group Co. LTD (Industry)
Collaborators: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY-2023-2-6-2
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Lung Injury
MeSH Terms: conditions — Lung Injury | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo control use saline (Placebo Comparator): saline is used as placebo in the placebo comparator group
  Interventions: Other: saline
- mesenchymal stem cells treatment (Experimental): Mesenchymal stem cell dose is 5×10*7/10ml and is transplanted by intravenous infusion. The cells are used once every three days and for three times.
  Interventions: Drug: mesenchymal stem cells

INTERVENTIONS:
Drug: mesenchymal stem cells — Mesenchymal stem cell dose is 5×10*7/10ml and is transplanted by intravenous infusion. The cells are used once every three days and for three times
  Other Names: KY-2023-2-6-2
  Arms: mesenchymal stem cells treatment
Other: saline — 10 ml saline is used as placebo once every three days and for three times
  Arms: placebo control use saline

SUMMARY:
The goal of this study is to conduct a prospective, double-blind, randomized placebo-controlled clinical trial to investigate the safety and efficacy of mesenchymal stem cells treatment for Lung injury caused by major infectious diseases.

DETAILED DESCRIPTION:
For patients with lung injury caused by major infectious diseases, conventional antiviral and anti-inflammatory treatments may not effectively improve lung function in the short term and may increase the risk of secondary infections. Therefore, in the clinical management of viral pneumonia, it is necessary to consider the lung tissue damage caused by acute viral replication and systemic immune stress, while also focusing on the subsequent lung functional impairment due to virus clearance-induced pulmonary fibrosis. Studies have shown that after peripheral intravenous administration of mesenchymal stem cells (MSCs), approximately 50% to 60% of the cells remain in the lung tissue within 1 hour, decreasing to around 30% after 3 hours. After 48 hours, MSCs tend to aggregate in the liver and spleen, and cell retention can still be detected 10 days later. MSCs aggregation in the lung tissue can secrete cell trophic factors such as keratinocyte growth factor (KGF), vascular endothelial growth factor (VEGF), and hepatocyte growth factor (HGF), promoting the regeneration of type II alveolar epithelial cells, improving the pulmonary microenvironment, and facilitating the repair of the alveolar epithelial barrier after ARDS injury.This study is intended to conduct a prospective, double-blind, randomized placebo-controlled clinical trial to investigate the safety and efficacy of mesenchymal stem cells treatment for Lung injury caused by major infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Understand and sign the informed consent form, comply with the relevant requirements of this study, and agree not to participate in other studies and not to receive other immunotherapy during the study participation;
3. meet the diagnosis of viral pneumonia and are in the advanced stage of disease: (1)The etiological diagnosis met any of the following criteria:

   ①Sars-cov-2 infection: Respiratory specimens (nasal/throat swabs or bronchial secretions/bronchoalveolar lavage fluid) were positive for Sars-cov-2 nucleic acid and/or antigen within 14 days;

   ②Adenovirus infection: positive for adenovirus nucleic acid and/or antigen in respiratory secretions or blood within 14 days;

   ③Influenza virus infection: positive respiratory secretions or blood for influenza virus nucleic acid and/or antigen within 14 days;

   ④Other respiratory virus antigens or nucleic acids were positive in respiratory secretions or blood within 14 days; (2)Imaging manifestations: chest X-ray or CT was consistent with the imaging features of viral pneumonia, manifested as multiple patchy shadows, ground glass shadows or consolidation in both lungs; (3)Respiratory System Indicators:Respiratory distress, respiratory rate (RR) ≥30 breaths/min at rest; In the resting state, oxygen saturation of finger pulse was ≤93% while breathing air; Oxygen and index (partial pressure of arterial oxygen/fraction of inspired oxygen) ≤300mmHg and > 200mmHg;
4. Invasive mechanical ventilation and vasopressor medications were not required.

Exclusion Criteria:

1. Patients tested active for HBV, HCV, HIV, or tuberculosis at the time of screening;
2. patients with solid tumors, leukemia or mental disorders;
3. The peripheral white blood cell count was still more than 12×109/L or less than 4×109/L after effective anti-infective treatment. Plasma C-reactive protein >2 times the upper limit of normal; Plasma procalcitonin >2 times the upper limit of normal;
4. There were severe complications or major organ complications: severe cardiovascular and cerebrovascular diseases: acute heart failure NYHAⅢ; uncontrolled myocarditis or valvular disease; malignant arrhythmia; incident (≤6 months) cardio-cerebrovascular events (myocardial infarction or stroke); previous chronic bronchitis, severe asthma, obstructive pulmonary emphysema, pulmonary fibrosis, and other diseases that require long-term oxygen therapy or affect daily activities; patients with acute renal failure (≥44.2 μmol/L daily increase in serum creatinine) or chronic renal insufficiency had serum creatinine ≥442 μmol/L; the liver function was markedly abnormal and ALT≥5×ULN; serum TBil≥10×ULN or daily increase ≥17.1 μmol/L; signs of bleeding, PTA≤ 40% (or INR≥1.5); severe anemia (Hb<60g/L), moderate or severe thrombocytopenia (PLT<60×109/L), and DIC; other conditions that the investigators thought might affect treatment effectiveness.
5. Unwillingness to sign informed consent forms;
6. Evidence of drug addiction within 6 months before trial entry;
7. Patients who are currently enrolled in other clinical trials and may violate this treatment regimen and observation indicators;
8. Unable or unwilling to provide informed consent or to comply with the study requirements;
9. Other serious conditions that may preclude the clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with side effects in MSCs treatment groups | 48 weeks
  Investiagte the number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after MSCs infusion.
High-resolution CT imaging | 2 weeks
  at week 2, evaluate high-resolution CT imaging changes in lung lesions and compare with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Fu sheng Wang, Dr, Principal Investigator — Beijing 302 Hospital
Locations (1):
- Beijing 302 Hospital, Beijing, China